CLINICAL TRIAL: NCT04359472
Title: The Collection and Application of Autologous Amniotic Fluid At Cesarean Delivery Closure - a Feasibility Study.
Brief Title: The Collection and Application of Autologous Amniotic Fluid At Cesarean Delivery Closure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recibio, Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEALOGIC-DUKE
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Related; Cesarean Wound Disruption; Cesarean Section; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Other): Collection and reapplication of amniotic fluid.
  Interventions: Device: Application of Autologous Amniotic Fluid

INTERVENTIONS:
Device: Application of Autologous Amniotic Fluid — Collection and reapplication of amniotic fluid at wound layers during a cesarean section.

SUMMARY:
The purpose of this study is to determine the feasibility of collecting amniotic fluid at delivery that will be immediately processed and then applied as a spray to the various layers of cesarean wound closure.

DETAILED DESCRIPTION:
This is a single-site, prospective pilot study involving the collection of amniotic fluid at cesarean delivery followed by the immediate processing and re-application to the closure among twenty women at term undergoing cesarean delivery at Duke University Hospital. The objective of the study is to determine the feasibility of collection and application of autologous amniotic fluid at cesarean delivery.

VISIT 1: Screening/Enrollment Visit:

Once informed consent is obtained, demographic information, as well as medical and surgical history will be obtained. A medical release form will also be signed so that in the event that the subject is seen outside the Duke Health system after delivery, the study team will be able to request pertinent medical records.

VISIT 2: Day of Surgery Visit:

At presentation for delivery, study team members will reconfirm eligibility criteria. Subjects will then undergo cesarean delivery as per standard care.

The Recibio kit includes the following supplies, all of which are packaged in a sterile kit and will be opened onto the sterile surgical field:

* Mucous trap
* Yankauer suction device
* Tubing to connect to wall suction
* 10 ml syringe
* 1 ml syringe
* Syringe spray applicator and spray tip with attached syringes - the spray device is included in sterile packaging and manufactured and distributed by Recibio, Inc. Ratio Applicator Kit, Ref # 2101 with an have FDA clearance via Class 1 exempt device FDA listing number D377967.

  10% calcium chloride vials will be provided separately. Vials will not be placed on the sterile field as it will likely not have sterile packaging. The calcium chloride solution will either be poured into a small sterile bowl so that it may be drawn up into the1 cc device syringe in a sterile manner OR drawn up into the device syringe directly by a member of the sterile surgical team while a member of the study team holds the non-sterile portion of the vial.

The sterile supplies will be placed on the surgical table and set up for use prior to the start of the cesarean section. The surgery will begin and be completed as part of standard of care.

Once the uterine incision has been made the following steps will be taken:

Following incision of the lower uterine segment, the amniotic sac will be opened with an amniotic perforator.

The Yankauer will be used to suction the amniotic fluid into the mucous trap as it escapes from the amniotic cavity.

After delivery of the newborn and placenta and the uterine incision closed, the amniotic fluid will be drawn from the mucous trap into the 10 ml syringe

The 10 mL syringe containing the amniotic fluid will then be observed for gross contamination (i.e. vernix, meconium-staining) and then attached to the spray device.

The 1 ml syringe containing 1 ml of 10% calcium chloride will then also be attached to the spray device via the second port (final concentration of 1% once sprayed).

The amniotic fluid-calcium chloride mixture will then be sprayed (1.5 to 2.0 ml) across the closed uterine incision and lower uterine segment.

Next the fascia will be closed and the fascial incision sprayed (1.5 to 2.0 ml).

Finally, the subcutaneous tissue will be closed and sprayed (1.5 to 2.0 ml) and then the skin will be closed and sprayed (1.5 to 2.0 ml).

A photo of the closed incision will be taken prior to the application of any bandages.

The incision will then be dressed as part of standard practice.

Any extra amniotic fluid will be kept and stored at -80 degrees in the Duke Reproductive Biology and Perinatal Research Laboratory for potential future research.

Since this study is testing product feasibility, only licensed investigators that are included as study personnel will be permitted to apply CeaLogic to the various tissue layers as described above.

Data elements regarding certain time points during surgery, use of the CeaLogic, and any complications will be recorded. These include, but are not limited to:

Procedure start time (incision time)

Time of uterine incision

Approximate volume of amniotic fluid collected

Description of amniotic fluid (color, presence/absence of vernix, blood, or meconium-staining)

Time that uterine closure is complete

Approximate spray volume to closed uterine incision

Approximate spray volume to closed abdominal fascia

Approximate spray volume to closed subcutaneous tissue

Approximate spray volume to closed skin

Procedure end time

Estimated blood loss

Type of skin closure

VISIT 3: Day of Discharge Visit:

The subject will receive routine post-operative care during the immediate post-operative period. Most cesarean section patients are discharged home on post-operative day 2 or 3. The following study activities will occur at this visit:

A photo of the incision site

Assessment of the incision site that includes presence of redness, swelling, induration, as well as pain at rest and with gentle pressure

The amount of pain medication used since delivery (non-steroidal anti-inflammatory agents and narcotics)

The patient will be provided with a memory aid to record pain level and any pain medications that she takes once she goes home.

An instruction form on how to complete the memory aid, as well as study team contact information, should the patient have questions or problems related to her incision.

Scheduling of the first follow up visit that will occur 6-8 days after surgery.

The study team will monitor the subject's medical record for vital signs and record any evidence of post-operative fever (maternal temperature greater than 38 degrees C its source, and action taken by the care team.

Documentation of any adverse events

VISIT 4: 1 Week Follow Up Visit:

Subjects will be seen at the Duke Perinatal Research Center approximately one week following her procedure (post-operative day 6-8).

At this visit the following study procedures will occur:

Photo of the wound

Assessment of the incision

Documentation of any signs or symptoms of infection

Review of the subject's memory aid for pain and pain medication

Documentation of any adverse events

Scheduling of the next study visit (approximately 4 weeks post-delivery)

VISIT 5: 4 Week Follow Up Visit:

Subjects will be seen during the routine postpartum clinic visit at approximately 4 weeks following delivery.

At this visit the following study procedures will occur:

Photo of the wound

Assessment of the incision

Documentation of any signs or symptoms of infection

Documentation of any adverse events

Review of the subject's memory aid for pain and pain medication

VISIT 6: Phone Call Follow Up Visit:

The subject will be contacted by telephone by a member of the study team approximately 6 weeks after delivery to determine if she had any wound complications since her last visit. If so, the subject's medical record will be reviewed to determine if there were any complications or treatment pertaining to her cesarean section incision. If the subject received this care outside of the Duke Health system, the signed medical records release will be sent to the applicable health care facility to request pertinent to be reviewed. An IRB-approved phone script will be used for this phone call. The subject will also be asked a series of questions pertaining to medication use, pain at the incision site, and activity level. Adverse events will be documented if they have occurred.

Unscheduled Study Visit:

If a study subject contacts the study team with concern for complications with her cesarean section wound, an unscheduled visit will be completed. This visit can happen anytime during the subject's participation(up to 30 days following the procedure where the procedure day is day 1), but after the CeaLogic has been applied.

During this visit, study staff will perform the following study procedures:

Photo of the wound

Assessment of the incision

Documentation of any signs or symptoms of infection

Documentation of adverse events

Review of medical record for any treatment actions taken related to the cesarean section wound

Product Use questionnaire:

In addition to the above study activities, each time a licensed investigator uses CeaLogic, they will be asked to complete a short questionnaire about their experience with using the device. No personal identifying information will be captured in this questionnaire. Information gathered from these questionnaires will be compiled and given to the sponsor for feedback and possible product improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant female age great than 18 years
2. Singleton gestation
3. Plan for cesarean delivery
4. Planned gestational age of at least weeks at the time of delivery
5. English speaking
6. Able to provide own informed consent
7. Intention of being available for entire study period and complete all relevant study procedures, including follow-up study visits and phone calls

Exclusion criteria at screening/enrollment:

1. Diabetes requiring therapy (type I or type II diabetes, gestational diabetes on medical therapy)
2. BMI greater than or equal to 40 kg/m2 at the time of enrollment
3. Placenta previa or placenta accreta
4. Prior bowel or urologic surgery (except un-ruptured appendectomy or uncomplicated cholecystectomy)
5. Multiple gestation
6. Previous history of postpartum hemorrhage requiring medical or surgical treatment
7. Known or suspected impairment of immunologic function including infection with HIV, hepatitis B or C
8. Known tobacco or drug use
9. Any condition which, in the opinion of the investigator, may pose a health risk to the subject or interfere with the evaluation of the study objectives
10. History of keloid formation

Exclusion criteria at time of surgery:

1. Labor at time of presentation to labor and delivery (regular, painful uterine contractions occurring every 5 minutes with evidence of cervical change)
2. Chorioamnionitis or other systemic infection at time of presentation for cesarean section, including evidence of lower abdominal skin infection (i.e. yeast, etc)
3. Need for urgent Cesarean section (examples include, but not limited to: non-reassuring fetal status (category II or III tracing), placental abruption, severe preeclampsia or eclampsia)
4. Rupture of membranes prior to the start of the surgery
5. Meconium-stained or blood-stained amniotic fluid
6. Experiences intraoperative hemorrhage requiring transfusion, disseminated-intravascular coagulopathy (DIC), or other medical or surgical condition during the delivery deemed by the investigator to pose a prohibitively high risk for surgical re-exploration or wound complication.
7. Who, in the investigator's opinion, would have any clinically significant condition that would impair the patient's ability to comply with the study procedures
8. Need for vertical skin incision
9. Intraoperative use of hemostatic agent (examples include FLOSEAL and AVIGUARD®)
10. Plan for use of staples at closure of the skin incision
11. Preeclampsia with severe features

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant female > 18 years old, single gestation, plan for cesarean delivery, planned gestational age > 37 weeks at the time of delivery, english speaking, able to provide own informed consent, intention of being available for entire study period
Enrollment: 20 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Collection and reapplication of autologous amniotic fluid | At time of delivery
  Feasibility of collection and reapplication of autologous amniotic fluid at the time of a cesarean delivery

SECONDARY OUTCOMES:
Cesarean Wound Complication | 6 weeks
  Cesarean wound disruption, infection, hematoma, seroma
Assessment of the Cesarean Wound | 4 weeks
  Assessment of would via validated cosmetic score using the Modified Hollander Score. This involves 6 incision attributes (e.g. step off boarders, contour irregularities, etc.) that are listed and a score of a 0 or 1 are given. A 0 means "No" the attribute does not exist which is good and a score of 1 means "Yes" the attribute does exist. After scoring all 6 attributes a 0 or a 1, the numbers are totaled with a being the best and 6 being the worst.
Pain Medication Use | 4 and 6 weeks
  Measure the patient's pain medication use
Pain Score | 4 and 6 weeks
  Measure the patient's pain using the visual analog scale (VAS). It is a scale from 1-10 where 1 is the lowest and 10 is the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gilner, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamilton BE, Martin JA, Osterman MJ. Births: Preliminary Data for 2015. Natl Vital Stat Rep. 2016 Jun;65(3):1-15. PMID 27309256
- [Background] Osterman MJ, Martin JA. Primary cesarean delivery rates, by state: results from the revised birth certificate, 2006-2012. Natl Vital Stat Rep. 2014 Jan;63(1):1-11. PMID 24461076
- [Background] American College of Obstetricians and Gynecologists (College); Society for Maternal-Fetal Medicine; Caughey AB, Cahill AG, Guise JM, Rouse DJ. Safe prevention of the primary cesarean delivery. Am J Obstet Gynecol. 2014 Mar;210(3):179-93. doi: 10.1016/j.ajog.2014.01.026. PMID 24565430
- [Background] Nisenblat V, Barak S, Griness OB, Degani S, Ohel G, Gonen R. Maternal complications associated with multiple cesarean deliveries. Obstet Gynecol. 2006 Jul;108(1):21-6. doi: 10.1097/01.AOG.0000222380.11069.11. PMID 16816051
- [Background] Faulk WP, Matthews R, Stevens PJ, Bennett JP, Burgos H, Hsi BL. Human amnion as an adjunct in wound healing. Lancet. 1980 May 31;1(8179):1156-8. doi: 10.1016/s0140-6736(80)91617-7. PMID 6155575
- [Background] Stock SJ, Kelly RW, Riley SC, Calder AA. Natural antimicrobial production by the amnion. Am J Obstet Gynecol. 2007 Mar;196(3):255.e1-6. doi: 10.1016/j.ajog.2006.10.908. PMID 17346544
- [Background] Brady C, Vang S, Christensen K, Isler J, Vollstedt K, Holt D. Use of autologous platelet gel in bariatric surgery. J Extra Corpor Technol. 2006 Jun;38(2):161-4. PMID 16921691
- [Background] Everts PA, Devilee RJ, Oosterbos CJ, Mahoney CB, Schattenkerk ME, Knape JT, van Zundert A. Autologous platelet gel and fibrin sealant enhance the efficacy of total knee arthroplasty: improved range of motion, decreased length of stay and a reduced incidence of arthrofibrosis. Knee Surg Sports Traumatol Arthrosc. 2007 Jul;15(7):888-94. doi: 10.1007/s00167-007-0296-x. Epub 2007 Feb 24. PMID 17323096
- [Background] Thiebes AL, Reddemann MA, Palmer J, Kneer R, Jockenhoevel S, Cornelissen CG. Flexible Endoscopic Spray Application of Respiratory Epithelial Cells as Platform Technology to Apply Cells in Tubular Organs. Tissue Eng Part C Methods. 2016 Apr;22(4):322-31. doi: 10.1089/ten.TEC.2015.0381. Epub 2016 Mar 18. PMID 26739252
- [Background] Trowbridge CC, Stammers AH, Woods E, Yen BR, Klayman M, Gilbert C. Use of platelet gel and its effects on infection in cardiac surgery. J Extra Corpor Technol. 2005 Dec;37(4):381-6. PMID 16524157